CLINICAL TRIAL: NCT04539171
Title: Effectiveness of a Group Intervention Through Education in Pain Neurophysiology and Exercise in Women With Fibromyalgia: a Quasi-experimental Study in Primary Care
Brief Title: Pain Neuroscience Education and Physical Exercise Program in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM001-BU-018
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia
Keywords: Central Nervous System Sensitization; Chronic pain; Fibromyalgia; Neuroscience; Patient education
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, controlled, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pain neuroscience education (Health education) and Physical exercise program: 6 weekly sessions (2 hours each), and a reminder session one month later
  Interventions: Other: Pain Neuroscience Education and Physical Exercise
- Control (No Intervention): Standard of care.

INTERVENTIONS:
Other: Pain Neuroscience Education and Physical Exercise — Patients assigned to the experimental group perform a PNE program consisting of seven sessions, with therapeutic PE. PNE is a health education intervention aims to provide up-to-date information on neuroscience advances in the field of chronic pain.
  Arms: Intervention

SUMMARY:
This study evaluates the effects of a pain neuroscience education (PNE) and physical exercise (PE) program in women with fibromyalgia. The intervention group receives PNE and PE program supervised by a physiotherapist and a Family Doctor and the control group standard care, in primary care.

DETAILED DESCRIPTION:
Objectives: To evaluate the effectiveness of a PNE and PE in patients with fibromyalgia (FM).

Design: Quasi-experimental, controlled, non-randomized study, in Primary Care facilities.

Intervention: 6 weekly sessions (2 hours each), and a reminder session one month later.

Main measurements: Compliance with FM criteria, assessed using the Widespread Pain Index (WPI) and the Severity of Symptoms (SS) questionnaires, impact of FM in daily life (Fibromyalgia Impact Questionnaire: FIQ) and quality of live. Assessments are made at baseline, one month following the 6th session, and during the 6- and 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women with FM (2010 American College of Rheumatology Diagnostic Criteria for fibromyalgia)
* Women ≥ 18 years
* Agree to participate in the study and sign informed consent.

Exclusion Criteria:

* Oncological pain
* Motor control alteration that prevents the execution of the planned PE program
* Patients with associated pathologies that make it impossible to perform physical exercise program
* Any disabling mental illness or intellectual deficit that prevents understanding the contents of PNE program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Fulfillment of diagnostic criteria for fibromyalgia | Change from baseline to 12 months follow-up
  2010 American College of Rheumatology Diagnostic Criteria for fibromyalgia: dichotomous variable (complies or does not comply). A patient satisfies diagnostic criteria for fibromyalgia if the following 3 conditions are met:
  1. Widespread pain index (WPI) ≥7 and symptom severity (SS) scale score ≥5 or WPI 3-6 and SS scale score ≥9.
  2. Symptoms have been present at a similar level for at least 3 months.
  3. The patient does not have a disorder that would otherwise explain the pain.
  WPI: number of areas in which the patient has had pain over the last week (score between 0 and 19), with 0 = fully active and 5 = dead).
  SS: sum of the severity of 3 symptoms (fatigue, waking unrefreshed, cognitive symptoms) plus the extent (severity) of somatic symptoms in general (final score between 0 and 12: higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Impact of fibromyalgia on daily life | Change from baseline to 12 months follow-up
  Evaluation of physical functionality, global impact and severity of symptoms: Fibromyalgia Impact Questionnaire (FIQ), which ranges from 0 to 100, with higher scores indicating worse outcome
Catastrophism | Change from baseline to 12 months follow-up
  Pain-related catastrophizing behaviours and cognitions of individuals: Pain Catastrophizing Scale (PCS), which ranges from 0 to 52, with higher scores indicating worse outcome
Anxiety | Change in score from baseline to 12 months follow-up
  Anxiety sub-scale of the Hospital Anxiety and Depression Scale (HAD), which ranges from 0 to 21, with higher scores indicating worse outcome
Depression | Change in score of both subscales from baseline to 12 months follow-up
  Depression sub-scale of the Hospital Anxiety and Depression Scale (HAD), which ranges from 0 to 21, with higher scores indicating worse outcome
Pain intensity | Change from baseline to 12 months follow-up
  Pain intensity sub-scale of the Brief Pain Questionnaire (BPI), which ranges between 0-40, with higher scores indicating worse outcome
Impact of pain in person's daily performance | Change from baseline to 12 months follow-up
  Pain impact sub-scale of the Brief Pain Questionnaire (BPI), which ranges between 0-70, with higher scores indicating worse outcome
Functional capacity | Change from baseline to 12 months follow-up
  Difficulty in performing activities of daily living: Health Assessment Questionnaire (HAQ), which ranges from 0 to 60, with higher scores indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Pilar San Teodoro-Blanco, MD, Principal Investigator — Gerencia de Atención Primaria de Burgos. Castilla-León Health Service (Sacyl)
Locations (1):
- Unidad de Fisioterapia Burgos Centro. GAP Burgos (Sacyl), Burgos, Spain

IPD SHARING:
Plan to Share IPD: Yes
We plan to share IPD, upon reasonable request, at the time the data be published. We will share all IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: At the time the study results are published.
Access Criteria: Upon reasonable request after an individualized evaluation of each request by the research team.

REFERENCES:
- [Derived] Areso-Boveda PB, Mambrillas-Varela J, Garcia-Gomez B, Moscosio-Cuevas JI, Gonzalez-Lama J, Arnaiz-Rodriguez E, Del Barco MBA, Teodoro-Blanco PS. Effectiveness of a group intervention using pain neuroscience education and exercise in women with fibromyalgia: a pragmatic controlled study in primary care. BMC Musculoskelet Disord. 2022 Apr 4;23(1):323. doi: 10.1186/s12891-022-05284-y. PMID 35379222